CLINICAL TRIAL: NCT07371481
Title: Results of Soft Tissue Grafting Around Implant in the Mandible Molar Area
Brief Title: CTG Versus Collagen Matrix for Peri-Implant Soft Tissue Augmentation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hanoi Medical University (Other)
Responsible Party: Principal Investigator, DUC NGUYEN MINH, DDS, Hanoi Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 01250159
Record Dates: First submitted 2026-01-19; First posted 2026-01-28 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Peri-implant Soft Tissue Deficiency; Insufficient Peri-implant Keratinized Tissue
Keywords: Peri-implant soft tissue augmentation; Connective tissue graft; Collagen matrix; Dental implant

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned in a 1:1 ratio to one of two parallel groups to receive either a connective tissue graft or a collagen matrix for peri-implant soft tissue augmentation, with no crossover between groups.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessment is performed by an independent examiner who is blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (2):
- Connective Tissue Graft (CTG) (Active Comparator): Peri-implant soft tissue augmentation using autogenous connective tissue graft.
  Interventions: Procedure: Connective Tissue Graft
- Collagen Matrix (Experimental): Peri-implant soft tissue augmentation using a collagen matrix.
  Interventions: Device: Collagen Matrix

INTERVENTIONS:
Device: Collagen Matrix — A porcine-derived collagen matrix is used for peri-implant soft tissue augmentation at the time of implant surgery, serving as a substitute for autogenous connective tissue grafting.
  Arms: Collagen Matrix
Procedure: Connective Tissue Graft — An autogenous connective tissue graft harvested from the patient is used for peri-implant soft tissue augmentation at the time of implant surgery.
  Arms: Connective Tissue Graft (CTG)

SUMMARY:
This randomized controlled trial compares two techniques for peri-implant soft tissue augmentation in the mandibular molar region: an autogenous connective tissue graft (CTG) and a collagen matrix. Adult patients requiring implant treatment with insufficient peri-implant soft tissue thickness will be randomly assigned to receive either CTG or a collagen matrix at the time of implant surgery.

The study aims to evaluate and compare changes in peri-implant soft tissue thickness, width of keratinized tissue, and soft tissue contour over a 9-month follow-up period, as well as the occurrence of postoperative complications. The results of this study will help determine whether a collagen matrix can provide clinical outcomes comparable to those of connective tissue grafting for peri-implant soft tissue augmentation.

DETAILED DESCRIPTION:
This randomized controlled trial is designed to compare two approaches for peri-implant soft tissue augmentation in the mandibular molar region: an autogenous connective tissue graft (CTG) and a collagen matrix. Adult patients with insufficient peri-implant soft tissue thickness will be enrolled and randomly allocated in a 1:1 ratio to receive either CTG or a collagen matrix at the time of implant surgery. Randomization will be performed using a block randomization method, and outcome assessment will be conducted by a blinded examiner.

Clinical and digital evaluations will be performed at predefined time points, including baseline and follow-up visits up to 9 months after surgery. Peri-implant soft tissue thickness, width of keratinized tissue, and soft tissue contour changes will be assessed using standardized clinical measurements and digital workflows based on intraoral scanning and cone-beam computed tomography where indicated. Postoperative healing and adverse events will be monitored throughout the follow-up period.

The study is conducted at a single academic center and is intended to provide comparative clinical data on the effectiveness and safety of collagen matrix versus connective tissue grafting for peri-implant soft tissue augmentation.

ELIGIBILITY:
Inclusion Criteria:

Adults aged 18 to 65 years.

Patients requiring dental implant treatment in the mandibular molar region.

Presence of insufficient peri-implant soft tissue thickness (< 2 mm).

Adequate general health to undergo minor oral surgery.

Ability and willingness to provide written informed consent and comply with study procedures.

Exclusion Criteria:

Systemic conditions or medications that may impair wound healing.

Heavy smoking (more than 10 cigarettes per day).

History of allergy or hypersensitivity to collagen-based materials.

Previous graft failure or complications at the intended implant site.

Loss of three or more adjacent teeth in the study area (excluding third molars).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change in peri-implant soft tissue thickness | Baseline (before surgery) to 9 months after surgery
  Change in peri-implant soft tissue thickness measured using standardized digital methods.

SECONDARY OUTCOMES:
Change in width of peri-implant keratinized tissue | Baseline to 9 months after surgery
  Change in the width of keratinized tissue around the implant measured clinically using standardized procedures.
Change in peri-implant marginal bone level | Baseline to 9 months after surgery
  Changes in marginal bone level assessed using cone-beam computed tomography where indicated.
Peri-implant clinical indices | Up to 9 months after surgery
  Assessment of peri-implant inflammation using standardized clinical indices.

OTHER OUTCOMES:
Postoperative complications and adverse events | Up to 9 months after surgery
  Incidence of postoperative complications, including soft tissue necrosis, infection, bleeding, implant failure, and other adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- Hanoi Medical University, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because the dataset contains sensitive clinical and imaging information, and data sharing was not included in the approved study protocol or informed consent.